CLINICAL TRIAL: NCT00470652
Title: Management of Acute Pain in the Emergency Department:Impact of a Computer-Assisted Support
Brief Title: Management of Acute Pain in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Societe Française de Medecine d'urgence (Other)
Responsible Party: Hugli Olivier, MD, MPH, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CIU-1
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Pain
Keywords: pain; Pain Measurement; Decision Making, Computer-Assisted; Informatics
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Pre-intervention patients admitted to our ED in the month prior to the intervention, before the 'computer-assisted decision support' is turned on (the intervention)
- 2: Short-term post-intervention cohort of patients admitted in the month following the initiation of the 'computer-assisted decision support' for pain management
  Interventions: Device: computer-assisted decision support
- 3: long-term post-intervention cohort of patients admitted on the 6th month following the initiation of the 'computer-assisted decision support' for pain management
  Interventions: Device: computer-assisted decision support

INTERVENTIONS:
Device: computer-assisted decision support — at the end of the pre-intervention period, the patient flow software was modified to open popup windows automatically when pain intensity was not documented or pain was not reevaluated within the recommended interval. The popup window also detailed appropriate pain treatment guidelines based on the documented pain intensity. In addition, the patient's icon in the flow software changed from black to red when pain intensity was >4/10. After a 10-day test period, the post-intervention data collection started.
  Other Names: informatics; information technology
  Groups: 2; 3

SUMMARY:
Oligoanalgesia1 has been widely recognized as an issue in emergency department.The purpose of our study is to assess the impact of the implementation of a computer-assisted support program to improve pain management in our ED.

DETAILED DESCRIPTION:
Inadequate pain management remains a major challenge for health care providers. Despite extensive research on the mechanisms of acute pain, identification of factors leading to poor pain management and development of evidence-based strategies, the transfer of this knowledge into effective clinical practices has been surprisingly slow. Oligoanalgesia1 has been widely recognized as an issue in emergency department (ED) patients. Acute pain is reported by 60-80% of ED inpatients but is frequently undertreated. Overall, an insufficient proportion of patients with acute pain receive any type of analgesia, and pain relief remains unsatisfactory. We showed that the implementation of guidelines improved pain management. However, rotation of the medical & nursing staff leads to the forgetting of guidelines. The purpose of our study is to assess the impact of the implementation of a computer-assisted support program to improve pain management in our ED.

ELIGIBILITY:
Inclusion Criteria:

Any patient admitted to our Emergency Department who is

* age > 16 years
* pain lasting =< 1 week or
* no pain on admission but pain during the ED stay

Exclusion Criteria:

* life-threatening condition requiring immediate admission in the OR or ICU
* no pain or pain lasting >1 week
* inability to give informed consent (intoxicated, psychiatric disorder, language problem, prisoner)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients discharged from our ED who either had pain on admission or suffered of a new pain while in our ED
Sampling Method: Non-Probability Sample
Enrollment: 631 (Actual)
Dates: Start 2007-05; Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier W Hugli, MD,MPH, Principal Investigator — Centre Hospitalier Universiataire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Decosterd I, Hugli O, Tamches E, Blanc C, Mouhsine E, Givel JC, Yersin B, Buclin T. Oligoanalgesia in the emergency department: short-term beneficial effects of an education program on acute pain. Ann Emerg Med. 2007 Oct;50(4):462-71. doi: 10.1016/j.annemergmed.2007.01.019. Epub 2007 Apr 18. PMID 17445949